CLINICAL TRIAL: NCT06405607
Title: Psilocybin vs Ketamine for Alcohol Use Disorder
Brief Title: Psilocybin or Ketamine for Alcohol Use Disorder: An Active Comparator Trial
Acronym: Psi or Ket
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Peggy C Nopoulos, Department Chair, Psychiatry, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202404714
Record Dates: First submitted 2024-05-02; First posted 2024-05-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence; Alcohol Abuse
Keywords: psychedelic; psilocybin; ketamine
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin Group (Arm 1) (Experimental): receives individual psychotherapy sessions plus a (30 mg) psilocybin session.
  Interventions: Drug: Psilocybin
- Ketamine Group (Arm 2) (Active Comparator): receives individual psychotherapy sessions plus a (0.75 mg/kg) ketamine session
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Psilocybin — 30 mg single dose
  Arms: Psilocybin Group (Arm 1)
Drug: Ketamine — 0.75 mg/kg weight-based single dose
  Arms: Ketamine Group (Arm 2)

SUMMARY:
This study will collect data that measures the effects of a psychedelic intervention on patients struggling with alcohol use disorder (AUD). The study design will be a double blind, randomized, active-comparator trial with two study arms. Subjects randomized to Arm 1 (n=40) will receive individual psychotherapy sessions plus a 30 mg dose of psilocybin. Arm 2 subjects (n=40) will receive individual psychotherapy sessions and a 0.75 mg/kg dose of ketamine.

ELIGIBILITY:
Inclusion criteria:

* Weight between 50kg and 150kg
* No known allergies to rescue medication
* For people capable of becoming pregnant, not pregnant and using contraception
* Not currently breastfeeding
* Meets criteria for DSM-V moderate to severe AUD.
* Have at least 4 heavy drinking days (5 or more standard drinks in a day) in the past 30 days.
* Not currently participating in formal treatment for AUD.
* No history of a of cerebrovascular accident, asthma, or significant alcohol withdrawal history
* No seizure disorder, coronary artery disease, heart failure, uncontrolled hypertension, insulin-dependent diabetes, pancreatitis, liver disease
* No hallucinogen or ketamine use in past 12 months
* No self-reported, personal, or familial history of specific psychotic disorders/episodes.
* No serious traumatic brain injury (TBI) in the past 2 years
* No substance use disorder other than AUD over the past 12 months
* If taking a GLP-1 agonist, stable dosage for past 3 months
* Family member/friend for pick-up, overnight post-drug session monitoring.
* No MRI contraindications

Exclusion Criteria:

Drug/medication assessment that yields: nonprescription medication use, nutritional supplement, or herbal supplement (except when approved by the study investigators), medically unstable, current medication use that has significant potential to interact with study drug (e.g., antidepressants, antipsychotics, psychostimulants, treatments for addictions, other dopaminergic or serotonergic agents, lithium, anticonvulsants, or benzodiazepines).

Psychiatric assessment that yields:1) history of severe suicide attempt, 2) current suicidality 3) first-degree relative with schizophrenia or schizoaffective disorder, 4) comorbid substance use disorder including cocaine, psychostimulant, or opioid use disorder within past 12 months 5) history of co-occurring psychotic episode/diagnosis including schizophrenia, schizoaffective disorder, schizophreniform, substance-induced psychosis, delusional disorder, or psychosis not otherwise specified, 6) high risk of adverse emotional or behavioral reaction based on the medical monitor's clinical evaluation that may also yield evidence of serious current stressors, a lack of meaningful social support, antisocial behavior, and/or serious personality disorders amongst other conditions.

Medical assessment that yields: serious ECG abnormalities (evidence of ischemia, myocardial infarction, QTc prolongation [QTc > .045]), serious abnormalities of complete blood count or chemistries, medical conditions that would preclude safe participation (significantly impaired liver function), or pregnancy.

MRI contraindication (pacemaker, etc.)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-Back for Alcohol to assess change | Weekly, over the course of 16 weeks
  Quantifies daily alcohol use

SECONDARY OUTCOMES:
T1rho | Twice (before intervention, post intervention): at week 1 and week 16
  Measures biological changes in the brain
Resting state fMRI | Twice (before intervention, post intervention):: at week 1 and week 16
  Measures biological changes in brain resting state global functional connectivity
EEG- signal complexity | Twice (before drug administration and at peak of drug experience) during week 3
  Measures electrical signal change

CONTACTS AND LOCATIONS:
Overall Officials: Peggy C Nopoulos, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States